CLINICAL TRIAL: NCT04597229
Title: Efficacy of Multigrain Supplementation in Type II Diabetes Mellitus: A Randomized Human Clinical Trial
Brief Title: Efficacy of Multigrain Supplementation in Type II Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Dr. Lee Lai Kuan, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LLKuan
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instant multigrain (Active Comparator): Oral instant multigrain supplement
  Interventions: Dietary Supplement: Instant multigrain supplement
- Standard care (No Intervention): Standard care without oral instant multigrain supplement

INTERVENTIONS:
Dietary Supplement: Instant multigrain supplement — A twice daily instant multigrain supplementation for 12 weeks
  Arms: Instant multigrain

SUMMARY:
The objective of this study is to evaluate the efficacy of instant multigrain supplementation on the glycemic status, cardiometabolic implications, oxidative stress and nutritional status in Type II DM patients.

DETAILED DESCRIPTION:
Type II DM is a highly prevalent and heterogeneous condition. New treatment modalities to complement existing interventions are therefore of great interest, including dietary interventions for primary prevention or as a possible therapeutic option that may confer beneﬁts beyond currently recommended conventional therapies. Hence, the present work aims to evaluate the efficacy of instant multigrain supplementation on the glycemic status, cardiometabolic implications, oxidative stress and nutritional status in Type II DM patients, as compare to standardized medication regimen.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the clinical trial are:

* Clinical diagnosis with Type II DM for at least 6 months' duration without clinically manifest complications (retinopathy, diabetic nephropathy, vascular diseases, foot ulcer - as diagnosed by the physician/recorded in database)
* Male or female
* Pharmacological treatment with metformin or insulin, or a combination of metformin and glibenclamide.
* Chronological age: 18 years and above
* Metabolically stable (current laboratory results for A1C 6.0-8.5%; or fasting plasma glucose 6.4-8.5 mmol/l)
* Not taking antioxidant/anti-inflammatory supplements (Example of antioxidant: vitamin C, vitamin E, grape seed extract, garlic capsule, ginkgo biloba) (Example of anti-inflammatory supplement: fish oil, curcumin extract, ginger extract, spirulina)

Exclusion Criteria:

* Having liver (chronic liver failure, cirrhosis, all types of hepatitis), kidney (chronic kidney disease, haemodialysis) or haematological (anaemia, thalassemia, haemophilia) disorders
* Active gastric/duodenal ulcer
* Psychiatric disease/mental retardation (bipolar disorder, depression, schizophrenia)
* Cancer (all types), and endocrine disorders (Cushing's disease, gigantism and hyperthyroidism).
* Alcohol and drug abuse (self-mentioned or as recorded in the medical card)
* Gestational Diabetes Mellitus
* Pregnancy/lactation
* Hormone replacement therapy (for at least 3 months prior to entering the study)
* Herbal remedies (any parts from the plants such as flowers, rhizome, seeds, roots, leaves, fruits, stems)
* Use of steroids, chemotherapy, immunosuppressant or radiotherapy.
* Vegetarian patient (pure vegan)
* Gluten intolerance
* Participations currently under another supplementary program

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Change of Glycated haemoglobin (HbA1c) | Baseline and 12 weeks
  Glycated hemoglobin (HbA1c) is measured in %
Change of fasting plasma glucose (FPG) | Baseline and 12 weeks
  Glycated hemoglobin (HbA1c) is measured in mmol/L
Change of fasting serum insulin | Baseline and 12 weeks
  Fasting serum insulin will be measured by radioimmunoassay kit

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Medical and Dental Institute (AMDI), Kepala Batas, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No